CLINICAL TRIAL: NCT04093557
Title: Validation of a Novel Clinical Prediction Scoring System for Improved Bowel Preparation Prior to Outpatient Colonoscopy
Brief Title: Improving Outpatient Colonoscopy Bowel Prep with the Orton Score
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough funding for research coordinator.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Steven Powell, MD, Associate Professor, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21825
Record Dates: First submitted 2019-09-13; First posted 2019-09-18 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-05

CONDITIONS: Colonic Polyp; Colon Cancer
Keywords: colonoscopy; bowel prep; screening
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients will be assessed for the most appropriate bowel preparation prior to colonoscopy (standard vs. extended) based on a novel scoring tool that accounts for various clinical conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Orton Score Cohort - High (Active Comparator): Patients will be scored using the "Orton Score," a novel clinical prediction tool to determine which patients are at risk for poor bowel preps and may benefit from an extended prep. If they score highly, they will receive an extended GoLytely bowel prep.
  Interventions: Other: Orton Score
- Prospective Orton Score Cohort - Low (Placebo Comparator): Patients will be scored using the "Orton Score," a novel clinical prediction tool to determine which patients are at risk for poor bowel preps and may benefit from an extended prep. If they do not score highly, they will receive a standard GoLytely (or Suprep) bowel prep.
  Interventions: Other: Orton Score
- Retrospective Cohort (before Orton Score) (Other)
  Interventions: Other: Typical Standard of Care

INTERVENTIONS:
Other: Orton Score — Significant a priori predictors of poor prep included: male gender, COPD, diabetes with end-organ damage, severe neurologic disease, constipation medication use, and tricyclic antidepressant use. Proprietary web-based weighted scoring model allows screening clinician to predict which bowel prep would be best for patient depending on which risk factors patients have.
  Arms: Orton Score Cohort - High; Prospective Orton Score Cohort - Low
Other: Typical Standard of Care — Clinician usual practice of prescribing bowel preps to patient
  Arms: Retrospective Cohort (before Orton Score)

SUMMARY:
Colonoscopy is a common endoscopic procedure which the UVA Gastroenterology & Hepatology department performs on a daily basis for both screening/surveillance and diagnostic/therapeutic intent. As a safety net hospital, the institution also offers open access colonoscopy as a means of allowing outside primary care and urgent care providers a way to have patients receive necessary endoscopy services. However, these patients are not all seen in clinic prior to their procedure but are all prescribed a specific bowel prep by a medical professional who screens the referrals.

Given that the patient population described above are often not well-known to UVA providers, they may be prescribed prep regimens that are not ideal for their comorbidities. Not infrequently, these patients show up to their colonoscopies with an inadequate bowel prep, leading to either cancelled or incomplete procedures, increased healthcare and personal financial costs (such as missed wages from taking off work), suboptimal endoscopy resource utilization, and delay in or missed polyp (or potentially cancer) detection.

The investigators seek to use a novel scoring system designed to predict patients at risk for suboptimal preps (and hence patients that would benefit from an extended prep) and apply it in uniform fashion to a patient population most at risk for suboptimal preps. Because obtaining written consent is not practical given that these patients may not be seen by a UVA provider prior to their endoscopic procedure, the investigators will plan to verbally consent via the telephone in an all-inclusive manner; there will be no randomization but rather the selection of prep to be determined by the novel scoring system. Subjects be prescribed either a standard split-dose GoLytely prep (or SuPrep) or an extended split-dose GoLytely prep. The investigators predict that utilizing this new system will lead to a decreased number of inadequate bowel preps and will increase polyp detection. The investigators will work with a UVA biostatistician to analyze the data and use Chi Square, student's T tests, and logistic regression models to assess significance and help validate the model.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older (up to 100 years)
* Referred for open access colonoscopy from an outside provider/UVA provider
* Able to provide informed consent

Exclusion Criteria:

* Prisoners

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Inadequate prep rate | Through study duration, approximately 1 year
  Percentage of colonoscopies where performing endoscopist rates the prep as inadequate for intended purpose (screening/surveillance)

SECONDARY OUTCOMES:
Adenoma detection rate (ADR) | Through study duration, approximately 1 year
  Percentage of colonoscopies with detection of at least 1 adenoma
Polyp burden | Through study duration, approximately 1 year
  Mean # of polyps found per colonoscopy
Advanced adenoma / adenocarcinoma detection rate | Through study duration, approximately 1 year
  Percentage of colonoscopies with detection of an adenoma with high-grade dysplasia, tubulovillous adenoma, or adenocarcinoma
Incomplete colonoscopy rate | Through study duration, approximately 1 year
  Percentage of colonoscopies that are unable to be completed secondary to inadequate prep or technical difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Powell, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson DA, Barkun AN, Cohen LB, Dominitz JA, Kaltenbach T, Martel M, Robertson DJ, Boland CR, Giardello FM, Lieberman DA, Levin TR, Rex DK; US Multi-Society Task Force on Colorectal Cancer. Optimizing adequacy of bowel cleansing for colonoscopy: recommendations from the US multi-society task force on colorectal cancer. Gastroenterology. 2014 Oct;147(4):903-24. doi: 10.1053/j.gastro.2014.07.002. No abstract available. PMID 25239068
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Sherer EA, Imler TD, Imperiale TF. The effect of colonoscopy preparation quality on adenoma detection rates. Gastrointest Endosc. 2012 Mar;75(3):545-53. doi: 10.1016/j.gie.2011.09.022. Epub 2011 Dec 3. PMID 22138085
- [Background] Lebwohl B, Kastrinos F, Glick M, Rosenbaum AJ, Wang T, Neugut AI. The impact of suboptimal bowel preparation on adenoma miss rates and the factors associated with early repeat colonoscopy. Gastrointest Endosc. 2011 Jun;73(6):1207-14. doi: 10.1016/j.gie.2011.01.051. Epub 2011 Apr 8. PMID 21481857
- [Background] Chokshi RV, Hovis CE, Hollander T, Early DS, Wang JS. Prevalence of missed adenomas in patients with inadequate bowel preparation on screening colonoscopy. Gastrointest Endosc. 2012 Jun;75(6):1197-203. doi: 10.1016/j.gie.2012.01.005. Epub 2012 Feb 28. PMID 22381531
- [Background] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020
- [Background] Khan MA, Piotrowski Z, Brown MD. Patient acceptance, convenience, and efficacy of single-dose versus split-dose colonoscopy bowel preparation. J Clin Gastroenterol. 2010 Apr;44(4):310-1. doi: 10.1097/MCG.0b013e3181c2c92a. No abstract available. PMID 19935082
- [Background] Marmo R, Rotondano G, Riccio G, Marone A, Bianco MA, Stroppa I, Caruso A, Pandolfo N, Sansone S, Gregorio E, D'Alvano G, Procaccio N, Capo P, Marmo C, Cipolletta L. Effective bowel cleansing before colonoscopy: a randomized study of split-dosage versus non-split dosage regimens of high-volume versus low-volume polyethylene glycol solutions. Gastrointest Endosc. 2010 Aug;72(2):313-20. doi: 10.1016/j.gie.2010.02.048. Epub 2010 Jun 19. PMID 20561621
- [Background] Eun CS, Han DS, Hyun YS, Bae JH, Park HS, Kim TY, Jeon YC, Sohn JH. The timing of bowel preparation is more important than the timing of colonoscopy in determining the quality of bowel cleansing. Dig Dis Sci. 2011 Feb;56(2):539-44. doi: 10.1007/s10620-010-1457-1. Epub 2010 Nov 2. PMID 21042853
- [Background] Siddiqui AA, Yang K, Spechler SJ, Cryer B, Davila R, Cipher D, Harford WV. Duration of the interval between the completion of bowel preparation and the start of colonoscopy predicts bowel-preparation quality. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):700-6. doi: 10.1016/j.gie.2008.09.047. PMID 19251013
- [Background] Ben-Horin S, Bar-Meir S, Avidan B. The outcome of a second preparation for colonoscopy after preparation failure in the first procedure. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):626-30. doi: 10.1016/j.gie.2008.08.027. PMID 19251002
- [Background] Gimeno-Garcia AZ, Hernandez G, Aldea A, Nicolas-Perez D, Jimenez A, Carrillo M, Felipe V, Alarcon-Fernandez O, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Moreno M, Ramos L, Quintero E. Comparison of Two Intensive Bowel Cleansing Regimens in Patients With Previous Poor Bowel Preparation: A Randomized Controlled Study. Am J Gastroenterol. 2017 Jun;112(6):951-958. doi: 10.1038/ajg.2017.53. Epub 2017 Mar 14. PMID 28291237
- [Background] ASGE Standards of Practice Committee; Saltzman JR, Cash BD, Pasha SF, Early DS, Muthusamy VR, Khashab MA, Chathadi KV, Fanelli RD, Chandrasekhara V, Lightdale JR, Fonkalsrud L, Shergill AK, Hwang JH, Decker GA, Jue TL, Sharaf R, Fisher DA, Evans JA, Foley K, Shaukat A, Eloubeidi MA, Faulx AL, Wang A, Acosta RD. Bowel preparation before colonoscopy. Gastrointest Endosc. 2015 Apr;81(4):781-94. doi: 10.1016/j.gie.2014.09.048. Epub 2015 Jan 14. No abstract available. PMID 25595062
- [Background] Chung YW, Han DS, Park KH, Kim KO, Park CH, Hahn T, Yoo KS, Park SH, Kim JH, Park CK. Patient factors predictive of inadequate bowel preparation using polyethylene glycol: a prospective study in Korea. J Clin Gastroenterol. 2009 May-Jun;43(5):448-52. doi: 10.1097/MCG.0b013e3181662442. PMID 18978506
- [Background] Mahmood S, Farooqui SM, Madhoun MF. Predictors of inadequate bowel preparation for colonoscopy: a systematic review and meta-analysis. Eur J Gastroenterol Hepatol. 2018 Aug;30(8):819-826. doi: 10.1097/MEG.0000000000001175. PMID 29847488
- [Background] Yadlapati R, Johnston ER, Gregory DL, Ciolino JD, Cooper A, Keswani RN. Predictors of Inadequate Inpatient Colonoscopy Preparation and Its Association with Hospital Length of Stay and Costs. Dig Dis Sci. 2015 Nov;60(11):3482-90. doi: 10.1007/s10620-015-3761-2. Epub 2015 Jun 21. PMID 26093612